CLINICAL TRIAL: NCT06694012
Title: Osaka Cardiometabolic Epidemiological Study: Ohtori Study Part 2
Acronym: OCES-2
Status: Recruiting | Type: Observational
Sponsor: Osaka Metropolitan University (Other)
Collaborators: The Ministry of Education, Culture, Sports, Science and Technology, Japan (Unknown)
Responsible Party: Principal Investigator, Tomoshige Hayashi, Professor, Osaka Metropolitan University
Other Study IDs: 2024-030; JP23K17444 (Other Grant/Funding Number: Japan Society for the Promotion of Science)
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Type 2 Diabetes; Diabetes Mellitus; Hypertension; Hyperglycemia; Hyperlipidemia; Dyslipidemia; Hyperuricemia or Gout; Hyperuricemia, Gout; Obesity; Obesity/Epidemiology; Obesity, Abdominal; Central Obesity; Visceral Fat; Chronic Kidney Disease(CKD); Atherosclerosis; Metabolic Syndrome; Hepatic Steatosis; Insulin Sensitivity/Resistance
Keywords: Type 2 Diabetes Mellitus; Hypertension; Hyperlipidemia; Dyslipidemia; Hyperuricemia; obesity; Abdominal obesity; Visceral fat; Visceral adiposity; Chronic Kidney Disease; Japanese; Metabolic Syndrome; Insulin Sensitivity; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hypertension; Hyperglycemia; Hyperlipidemias; Dyslipidemias; Hyperuricemia; Gout; Obesity; Obesity, Abdominal; Renal Insufficiency, Chronic; Atherosclerosis; Metabolic Syndrome; Fatty Liver; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples stored in serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the relationship between body fat distribution measured by CT scan and related risk factors with the risk of incident metabolic and cardiovascular disease in a prospective cohort study of Japanese men and women. The investigators will also investigate novel risk factors for metabolic and cardiovascular disease using molecular weight-based metallomics analysis.

DETAILED DESCRIPTION:
Obesity is on the rise worldwide and is the most important risk factor for lifestyle-related diseases, including type 2 diabetes, hypertension, dyslipidemia, metabolic syndrome, ischemic heart disease, cerebrovascular disease, hyperuricemia, and chronic kidney disease. In addition, it has been reported that the distribution of fat is more important than the total amount of fat in the body, and the importance of visceral fat accumulation in the abdomen has been reported.

Although visceral fat accumulation and insulin resistance have been reported to be important upstream factors in the development of lifestyle-related diseases, the major target organs of insulin are not only adipose tissue, but also extremely important tissues such as muscle and liver, and ectopic fat accumulation in these tissues has attracted attention. However, there are few prospective cohort studies that have evaluated fat accumulation in adipose tissue, liver, and muscle simultaneously.

It has been reported that Japanese people have more visceral fat than Caucasians in the United States, even at the same body mass index level, and are at high risk for type 2 diabetes, so research on Japanese people is of great importance.

In addition, the role of trace elements in the body is attracting attention. In this cohort study, the investigators will also examine the relationship between trace elements in the body and the prevalence and incidence of lifestyle-related diseases.

The purpose of this study is to establish a prospective cohort study that evaluates visceral fat, subcutaneous fat, intrahepatic fat accumulation, and intramuscular fat using computed tomography imaging and to clarify the relationship with lifestyle-related diseases such as type 2 diabetes, hypertension, dyslipidemia, metabolic syndrome, ischemic heart disease, cerebrovascular disease, hyperuricemia, and chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Women who may be pregnant

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Japanese men and women aged 20 years or older who plan to undergo a health examination at the Ohtori Health Promotion Center in Sakai, Osaka, Japan, after November 2024 and who agree to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2050-03-31 (Estimated); Study Completion 2050-03-31 (Estimated)

PRIMARY OUTCOMES:
Type 2 diabetes is diagnosed based on the results of a fasting blood glucose test and medication history. | Investigators plan to conduct follow-up examinations at intervals of one to two years.
  Type 2 diabetes at baseline and follow-up examination is defined if the fasting plasma glucose level is ≥126 mg/dL, if the A1c level is ≥6.5%, or if the participant is taking medications or using injectables such as insulin to lower blood glucose levels at the baseline and follow-up examinations.
Hypertension is diagnosed based on the results of blood pressure measurement and medication history. | Investigators plan to conduct follow-up examinations at intervals of one to two years. plan to conduct follow-up examinations at intervals of one to two years.
  Hypertension is diagnosed if the systolic blood pressure is ≥140 mmHg, the diastolic blood pressure is ≥90 mmHg, or the participant is taking antihypertensive medications.
Dyslipidemia is diagnosed based on the National Cholesterol Education Program (NCEP) Adult Treatment Panel III guidelines. | Investigators plan to conduct follow-up examinations at intervals of one to two years. plan to conduct follow-up examinations at intervals of one to two years.
  Dyslipidemia is diagnosed based on the following criteria:Total cholesterol: ≥200 mg/dL (high); LDL cholesterol: ≥130 mg/dL (high); HDL cholesterol: <40 mg/dL (low in men), <50 mg/dL (low in women); or triglycerides: ≥150 mg/dL (high).
Metabolic syndrome is diagnosed based on the Joint Interim Statement published in Circulation. 2009 Oct 20;120(16):1640-5. | Investigators plan to conduct follow-up examinations at intervals of one to two years. plan to conduct follow-up examinations at intervals of one to two years.
  An individual is diagnosed with metabolic syndrome if they meet three or more of the following criteria:
  1. Abdominal obesity (waist circumference):
     Men: ≥90 cm Women: ≥80 cm
  2. Elevated triglycerides:
     Triglycerides ≥150 mg/dL, or receiving treatment for elevated triglycerides.
  3. Low HDL cholesterol:
     Men: <40 mg/dL Women: <50 mg/dL, or receiving treatment for low HDL cholesterol.
  4. Elevated blood pressure:
     Systolic blood pressure ≥130 mmHg, diastolic blood pressure ≥85 mmHg, or receiving antihypertensive treatment.
  5. Elevated fasting blood glucose:
  Fasting blood glucose ≥100 mg/dL, or receiving treatment for elevated blood glucose.
Hyperuricemia is defined based on fasting serum uric acid levels and the use of oral medication. | Investigators plan to conduct follow-up examinations at intervals of one to two years. plan to conduct follow-up examinations at intervals of one to two years.
  Hyperuricemia is diagnosed if the fasting serum uric acid levels is >7.0 mg/dL for men, >7.0 mg/dL for women, or if the participant is taking uric acid-lowering medication.
Low eGFR was define based on the Modification of Diet in Renal Disease study equation for Japanese. | Investigators plan to conduct follow-up examinations at intervals of one to two years. plan to conduct follow-up examinations at intervals of one to two years.
  Low eGFR was defined if eGFR was less than 60 mL/min/1.73 m², regardless of the presence of proteinuria.

CONTACTS AND LOCATIONS:
Overall Officials: Tomoshige Hayashi, MD, PhD, Principal Investigator — Osaka Metropolitan University
Locations (1):
- The Ohtori Health Promotion Center, Sakai, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No